CLINICAL TRIAL: NCT06090071
Title: A Phase 4, Single-Site Study Assessing Improvement of Skin Discoloration and Texture With Combination Treatment of Novel Moisturizer and Non-Ablative Laser Treatment Inclusive of Fitzpatrick Skin Types I-VI and Asian Descent
Brief Title: Trial Evaluating Both Tolerability and Improvement for Signs of Facial Photoaging, Discoloration, and Texture in Adult Females of All Skin Types by Combining a Placebo Moisturizer and Non-ablative Laser.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Austin Institute for Clinical Research (Network)
Collaborators: SkinCeuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDCR-000297
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Photoaging
Keywords: facial dyschromia

STUDY DESIGN:
Intervention Model Description: Split-Face study design. Phyto A+ Brightening Treatment and placebo moisturizer will be randomized regardless of Fitzpatrick Skin Type (FST). Subjects will be assigned to a laser treatment based on their Fitzpatrick Skin Type, as determined by the Investigator. Subjects with FST I-III will receive the Sciton laser procedure. Subjects with FST IV-VI will receive LaseMD laser procedure. Half of the face will be treated with Phyto A+ Brightening Treatment and assigned laser treatment. The other half of the face will be treated with placebo moisturizer and assigned laser treatment.
Who Masked: Participant, Investigator
Masking Description: Phyto A+ Brightening Treatment and placebo moisturizer will be labeled as Study Product A or Study Product B. Subjects, delegated site staff, or investigators will not know which product is applied to either side of the face.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Phyto A+ Brightening Treatment (Active Comparator): Phyto A+ Brightening Treatment is a serum comprised of a soothing botanical blend matched with a keratolytic (3% azeleic acid), 2.5% niacinamide, a brightening compound (2 % α-arbutin), and botanical extracts. Product will be topically applied to the assigned side of the face, either left or right side, at Day 0, Day 14, Day 28, Day 42, Day 70, and Day 98.
  Interventions: Device: LaseMD Laser; Device: Sciton Laser; Drug: Phyto A+ Brightening Treatment
- Placebo Moisturizer (Placebo Comparator): Placebo Moisturizer will be topically applied to the assigned side of the face, either left or right side, at Day 0, Day 14, Day 28, Day 42, Day 70, and Day 98.
  Interventions: Device: LaseMD Laser; Device: Sciton Laser; Drug: Phyto A+ Brightening Treatment

INTERVENTIONS:
Device: LaseMD Laser — The non-ablative fractional 1,927nm Thulium laser will be used in this study. This FDA-approved laser is an innovative device addressing as well as medical as aesthetic and cosmetic indications. The system allows nearly pain free treatments with depth of 200 μm setting multiple microbeams. The stratum corneum stays intact despite superficial ruptures, coagulation zones appear only in the underlying layers of the skin.
Device: Sciton Laser — The Sciton Laser uses Broadband light (BBL), also known as intense pulse light, a commonly available and popular treatment to rejuvenate the skin. BBL uses a broad band of noncoherent light waves, ranging from 560 to 1,200 nm, that are absorbed by a number of components in the skin, leading to a reduction in dyschromia, background erythema, telangiectasia, and an increase in collagen production resulting in amelioration of fine lines.
Drug: Phyto A+ Brightening Treatment — Phyto A+ Brightening Treatment is a serum comprised of a soothing botanical blend matched with a keratolytic (3% azeleic acid), 2.5% niacinamide, a brightening compound (2 % α-arbutin), and botanical extracts

SUMMARY:
This is a phase 4 trial evaluating the clinical effect of combining a placebo moisturizer and non-ablative laser to improve procedural outcomes in patients with facial dyschromia. This study's objective is to evaluate both the tolerability and improvement in signs of photoaging for a placebo moisturizer used in combination with a non-ablative laser. Physician assessments, patient reported outcomes, and digital photos will be captured.

DETAILED DESCRIPTION:
A single-site study that will enroll approximately 40 healthy female subjects, 25 to 70 years old, who meet all the inclusion and none of the exclusion criteria will be eligible to participate in this study subjects. The study population will include 15 patients with Fitzpatrick Skin Type I-III, 10 patients with Fitzpatrick Skin Type IV-VI, and 15 patients of Asian descent. The study duration is 14 weeks (98 days) including 6 study visits. This study's objective is to evaluate both the tolerability and improvement in signs of photoaging for a placebo moisturizer used in combination with a non-ablative laser. Physician assessments, patient reported outcomes, and digital photos will be captured. Clinical Efficacy endpoints will be evaluated at Day 0 (Baseline), Day 14 (Procedure), Day 28, Day 42, Day 70, and Day 98. Clinical efficacy assessments include Live Clinical Investigator Assessment, Redness, Skin Clarity, Appearance of Pores, Skin Texture/Smoothness (Visual), Skin Texture/Smoothness (Tactile), Hyperpigmentation, Skin Tone Evenness, Radiance/Brightness and Overall Healthy Appearance of Skin/Overall Skin Quality. The Modified Griffith's Scale will also be included. Tolerance endpoints will be evaluated at Day 0, Day 14 (Procedure), Day 28, Day 42, Day 70, and Day 98 including Objective Tolerance Evaluation and Subject Self-Assessment Tolerance. Instrumentation will be captured at Day 0 (Baseline), Day 14 (Procedure), Day 28, Day 42, Day 70, and Day 98 by VISIA Imaging Procedures (Canfield Imaging Systems) Before/After Photos. Subject Self-assessment Improvement and Product Use will be evaluated at Day 14 (Procedure), Day 28, Day 42, Day 70, and Day 98.

All participating subjects will receive the Phyto A+ Brightening Treatment (Pre-Treatment) and placebo prior to receiving the Fitzpatrick Skin Type (FST) appropriate laser treatment, as determined by the Investigator. On Day 14 subjects will be treated with a non-ablative based device treatment, Sciton or LaseMD. The LaseMD Laser allows nearly pain free treatments with depth of 200 μm setting multiple microbeams. The stratum corneum stays intact despite superficial ruptures, coagulation zones appear only in the underlying layers of the skin. The Sciton Laser uses a broad band of noncoherent light waves that are absorbed by a number of components in the skin, leading to a reduction in dyschromia, background erythema, telangiectasia, and an increase in collagen production resulting in amelioration of fine lines.

The occurrence of an adverse event (AE) or serious adverse event (SAE) may come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by a study monitor. All AEs including local and systemic reactions not meeting the criteria for SAEs will be captured on the appropriate case report form (CRF). Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of the event. All AEs occurring while on study must be documented appropriately regardless of relationship. Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode. Site staff will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit. All AE/SAEs will be followed for outcome information until resolution or stabilization. In accordance with the standard operating procedures and policies of the local Institutional Review Board (IRB), the site investigator will report SAEs to the IRB.

Protocol deviations will be captured and recorded when the subject, Investigator, or Sponsor fails to adhere to significant protocol requirements affecting the inclusion, exclusion, subject safety and primary endpoint criteria. Protocol deviations for this study include, but are not limited to, failure to meet inclusion/exclusion criteria. All significant protocol deviations will be reported to the IRB, in accordance with the standard operating procedures and policies of the local Institutional Review Board (IRB).

A subject may be discontinued from study treatment at any time if the subject, the Investigator, or the Sponsor feels that it is not in the subject's best interest to continue. The following possible reasons for study treatment discontinuation include Subject withdrawal of consent, Subject is not compliant with study procedures, Adverse event that in the opinion of the investigator would be in the best interest of the subject to discontinue study treatment, Protocol violation requiring discontinuation of study treatment, Lost to follow-up, Sponsor request for early termination of study, and Positive pregnancy test. If a subject is withdrawn from treatment due to an Adverse Event, the subject will be followed and treated by the Investigator until the abnormal parameter or symptom has resolved or stabilized. All subjects who discontinue study treatment should come in for an early discontinuation visit as soon as possible and then should be encouraged to complete all remaining scheduled visits and procedures. All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice. Reasonable attempts will be made by the Investigator to provide a reason for subject withdrawals. The reason for the subject's withdrawal from the study will be specified in the subject's source documents.

The investigational site will perform internal quality management of study conduct, data collection, documentation and completion. An individualized quality management plan will describe the site's quality management. Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution. Following written Standard Operating Procedures (SOPs), the monitors will verify that the clinical trial is conducted and data are generated and biological specimens are collected, documented (recorded), and reported in compliance with the protocol, International Conference on Harmonization Good Clinical Practice (ICH GCP), and applicable regulatory requirements (e.g., Good Laboratory Practices (GLP), Good Manufacturing Practices (GMP)). The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

The determined sample size is 40 subjects (N=15 Fitzpatrick I-III, N=10 Fitzpatrick IV-VI, N=15 Asian descent). The per-protocol (PP) population will be the primary population for all statistical analyses. The PP population will include all subjects who received treatment and completed the study in general accordance with the protocol. Only the data of completing subjects will be analyzed. Subjects may be removed from the analysis in the case of an AE, SAE, noncompliance, or Investigator decision. The reason for any subject(s) excluded from an analysis population will be documented and included in the study report. Demographic data and baseline characteristics, including age, sex, race, ethnicity, skin type (normal, oily, dry, combination), self-perceived sensitive skin (yes/no), and Fitzpatrick skin type, will be summarized according to the analysis population. For continuous variables, descriptive statistics including number of subjects (N), mean, median, standard deviation (SD), minimum (MIN), and maximum (MAX) values will be presented. For categorical variables, the frequency and percentage of each category will be provided. A descriptive statistical summary will be provided for all efficacy grading parameters and tolerability evaluation parameters. The descriptive statistical summary includes the N, mean, median, SD, MIN, and MAX of scores/values at all applicable time points for both sides of the face. The statistical analysis baseline will be Day 0. Mean of the change from baseline (defined as post-baseline value minus baseline value) will be estimated at applicable post-baseline time points. The null hypothesis, that the mean change from baseline is zero, will be tested using methods described in the Statistical Analysis Plan table. For efficacy grading parameters, a Shapiro-Wilk test will be used to test for normality of the baseline data (T0) and the change from baseline data (Tn-T0) at post-baseline time points at significance level alpha ≤0.05. When data passes normality (all normality of the distributions is confirmed for the same parameter), a parametric test will be used to test the null hypothesis that the mean change from baseline is zero. When data fails normality (if one or more normality of the distributions for the same parameter is rejected), a non-parametric test will be used. The following will be calculated and reported for each evaluation parameter at applicable post-baseline time point(s): Percent mean change from baseline = (time point mean score - baseline mean score) x 100. For applicable parameters, comparisons between the treated and untreated sides will be made in terms of changes from baseline. The null hypothesis, that the mean change from baseline is equal between the 2 sides at post-baseline time points, will be tested using methods described in the Statistical Analysis Plan Table. Questionnaire response options will be in the form of a 9-point semi-structured scale, ranging from 1 to 9, where the score of 1 will be the most negative/unfavorable rating and the score of 9 will be the most positive/favorable rating the product can receive (the scale will also include a mid-point label "neither agree nor disagree"). Responses obtained for each question will be tested for normality using a Shapiro-Wilk test at significance level alpha ≤ 0.05, and if the data passes normality testing, mean scores will be used. Responses that are not normally distributed will be assessed using the median response. The percentage of ratings from 6 to 9 will be reported. For questionnaire data, change from baseline analysis and comparison between treatments will be performed in the same way as for efficacy parameters. Any subjects who miss a questionnaire time point will be excluded from questionnaire analysis. In the report appendices, raw data will be listed by subject. Data frequency and percentage will be presented for questionnaires and tolerability evaluations. These tables will also be sent to the Sponsor at the indicated interim data time points. Medians, means and percentage values will be reported to 1 decimal place (0.0) for all questionnaire data. All statistical tests will be 2-sided at significance level alpha=0.05 unless specified otherwise. P values will be reported to 3 decimal places (0.000). No multiple testing corrections will be considered in the study. Statistical analyses are performed using SAS software version 9.4 (SAS Statistical Institute). The statistical results will be sent to the Sponsor along with raw data in a Microsoft Excel document at completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects aged between 25 and 70 years, all skin types included
2. Symmetrical photoaging
3. No known medical conditions that, in the Investigator's opinion may interfere with study participation
4. Willingness to cooperate and participate by following study requirements
5. Female subjects of childbearing potential must be willing to use appropriate contraception method(s)
6. Individuals must sign an informed consent and a photography consent

Exclusion Criteria:

1. Subjects that are being treated for cancer or have a history of facial skin cancer on the test areas
2. Subjects with sunburn, moderate to pronounced suntan, pronounced asymmetric skin aging, tattoos, scars or other disfiguration, dilated vessels or other conditions on the test area that might include the test results
3. Subjects currently taking certain medications which in the opinion of the Investigator(s) may interfere with the study. This includes but is not limited to routine high dosage use of anti-inflammatory drugs (aspirin, ibuprofen, corticosteroids [steroid nose drops, inhalers and/or eye drops are permitted]), and immunosuppessive drugs
4. Subjects with self-reported, uncontrolled systemic disease which, in the opinion of the Investigator, may hinder either the subject's ability to perform all responsibilities of the trial or the Investigator's ability to perform assessments
5. Women known to be pregnant, nursing or planning to become pregnant
6. Subjects participating in other facial clinical studies
7. Subjects who have routinely used an alpha-hydroxy-acid (AHA) or a beta-hydroxy-acid (BHA) containing product within two weeks or Retin-A, Retin-A Micro, Renova, Differin, Avita, Tazorac, or Soriatane within 8 weeks of the study start or have taken Isotretinoin within one year of the study start.
8. Subjects who have used Retinol in the last 4 weeks
9. Subjects with current flaring severe inflammatory acne
10. Subjects who have had ablative laser treatments, microneedling, and/or chemical peels or dermabrasion within the last six months
11. Subjects who have had botulinum type-A toxin (e.g. Botox®, Daxxify®, Dysport®, Jeaveau®, or Xeomin®) within the last 6 months
12. Subjects who have had dermal filler injections within the last 12 months
13. Subjects who have had non-ablative laser treatments or IPL within the last 3 months
14. Subjects with known allergies to skin treatment products or cosmetics, toiletries, and/or topical drugs
15. Subjects currently using topically applied prescription medications on the face

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Change in facial dyschromia | Change from Baseline to Day 98
  Measured by Live Clinical Investigator Assessment including, Skin Clarity, Appearance of Pores, Skin Texture/Smoothness (Visual), Skin Texture/Smoothness (Tactile), Hyperpigmentation, Skin Tone Evenness, Radiance/Brightness and Overall Healthy Appearance of Skin/Overall Skin Quality, and Tolerance Evaluation. Local cutaneous tolerability will be evaluated by assessing the signs of erythema, dryness, and scaling and by subject reporting of the degree of burning, stinging, and itching. Local cutaneous tolerability will all be measured with the parameters of 0 = none, 1 = mild, 2 = moderate, 3 = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, MBA, Principal Investigator — Austin Institute for Clinical Research
Locations (1):
- Austin Institute for Clinical Research, Inc., Pflugerville, Texas, United States